CLINICAL TRIAL: NCT04935203
Title: Can we Prime Sustainable Food Choice? A Mix-methods Study
Brief Title: Consumers' Emotional Reaction to Sustainability Cue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Qiuyan Liao, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201901231sv_b
Record Dates: First submitted 2021-06-07; First posted 2021-06-22 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Sustainable Food Consumption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control message group (No Intervention): Participants will not receive the priming manipulation.
- Health benefits priming group (Experimental): Participants will be cueing with health benefits by asking to do a word-search exercise beginning with: "In the following, please choose words/statements that can indicate that having a healthy and sustainable diet can have health benefits, such as..."
  Interventions: Behavioral: Priming intervention
- Environmental benefits priming group (Experimental): Participants will be cueing with environmental benefits by asking to do a word-search exercise beginning with: "In the following, please choose words/statements that can indicate that having a healthy and sustainable diet can have environmental benefits, such as..."
  Interventions: Behavioral: Priming intervention
- Environmental and health co-benefits priming group (Experimental): Participants will be cueing with environmental and health co-benefits by asking to do a word-search exercise beginning with: "In the following, please choose words/statements that can indicate that having a healthy and sustainable diet can have both benefits for health and the environment, such as..."
  Interventions: Behavioral: Priming intervention

INTERVENTIONS:
Behavioral: Priming intervention — The priming manipulation will be embedded in one computerized experiment to test the effect of three priming interventions on people's emotional reaction and their subsequent sustainable food selection. The priming conditions include priming with health benefits, environment benefits, and co-benefits of having sustainable diets, respectively. The cueing manipulation will be achieved by asking participants to complete a word-search exercise. Brief introduction will be provided to guide participants to choose words/statements that can indicate having a health and sustainable diet can have one of the three benefits: health benefits, environmental benefits or both benefits. The exercise will take ~2 min.
  Arms: Environmental and health co-benefits priming group; Environmental benefits priming group; Health benefits priming group

SUMMARY:
This will be a randomized control trial (RCT) to examine whether the three priming interventions (health priming, environmental sustainability priming, and co-benefits priming) work to change consumers' sustainable food choice through their effects on changing consumers' emotional reaction when seeing foods with cues of environmental sustainability, which will be indicated by measuring consumers' facial expression, eye movement and pupil dilation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be aged 18 years or above
* Subjects should be Hong Kong residents
* Subjects should be able to read Chinese

Exclusion Criteria:

* Subjects who have vegan or vegetarian diets will be excluded
* Subjects who have to follow special diets due to illnesses will be excluded
* Subjects domestic helpers will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Participants' choice of sustainable foods | Immediately after they are exposed to priming manipulation
  Measure name: Participants' food choice for sustainable food
  Measure tool: E-prime
  Measure process: During the computerized task, participants will examine a series of food products. Subsequently participants will be directed to simulated webpage for online shopping with all the foods they have examined available and they are required to buy three products they like most with the available budget provided.
  Measure units: Participants' actual food choice, whether they prefer choosing more sustainable food.
Participants' facial expression | Immediately after they are exposed to priming manipulation
  Measure name: Participants' facial expression measured by pupil diameters
  Measure tool: E-prime with Tobii Pro eye trackers
  Measure units: Pupil diameters will be used to compare difference when participants view the less or more sustainable foods. The larger pupillary variations is an indicator of interest in the products.
Participants' eye movement data | Immediately after they are exposed to priming manipulation
  Measure name: Participants' eye movement data
  Measure tool: E-prime with Tobii Pro eye trackers
  Measure units: Count frequency of looking at the environmentally friendly logo for each food category. Greater number indicates greater degree of attention and interest.

SECONDARY OUTCOMES:
Social orientation value | Immediately after they complete the computerized task with priming manipulation
  Measure name: Social Orientation Value (SVO)
  Measure tool: survey questionnaire
  Measure units: Participants will be classified as prosocial, individualistic, or competitive if they made at least six or more choices consistent with one of the orientations.
Pro-environmental values | Immediately after they complete the computerized task with priming manipulation
  Measure name: New Environmental Paradigm (a reduced 6-items version)
  Measure tool: Survey questionnaire
  Measure unit: All the responses will be measured on a 5-point agreement scale. Greater aggregated score indicates greater environmental concern.

CONTACTS AND LOCATIONS:
Locations (1):
- Jockey Club Tower, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request from PI.